CLINICAL TRIAL: NCT05218070
Title: Safety and Immunogenicity Study of EgyVax Vaccine Candidate for Prophylaxis of Severe Acute Respiratory Syndrome (SARS) - Coronavirus 2 (CoV-2) Infection (COVID-19)
Brief Title: Safety and Immunogenicity Study of EgyVax Vaccine Candidate for Prophylaxis of COVID-19 Infection
Acronym: Sphinx
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eva Pharma (Industry)
Collaborators: Veterinary Serum & Vaccine Research Institute (VSVRI), Egypt (Unknown); The Supreme Council of University Hospitals, Egypt (Unknown); Ministry of Higher Education and Scientific Research, Egypt (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: SPHINX22122020
Record Dates: First submitted 2022-01-25; First posted 2022-02-01 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose Vaccine (Experimental): 35 mcg dose for both vaccinations at day 0 and day 14 (low dose, 15 subjects)
  Interventions: Drug: EgyVax Vaccine Candidate
- High Dose Vaccine (Experimental): 70 mcg dose for both vaccinations at day 0 and day 14 (high dose, 15 subjects)
  Interventions: Drug: EgyVax Vaccine Candidate
- Placebo (Placebo Comparator): Placebo for both injections at day 0 and day 14 (Placebo, 15 subjects)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EgyVax Vaccine Candidate — EgyVax Inactivated SARS-CoV-2 vaccine candidate, equivalent to 70 mcg inactivated SARS-CoV-2 total protein. Alum adjuvant 2% 50 µl (equivalent to 0.5 mg AlOH). Equivalent volume of Saline 0.9% to each vaccine dose. Each vial contains 0.5 ml representing one dose 70 mcg of inactivated SARS-CoV-2 virus with alum adjuvant or two doses of 35 mcg of inactivated SARS-CoV-2 virus with alum adjuvant
  Arms: High Dose Vaccine; Low Dose Vaccine
Drug: Placebo — 0.5ml Saline (0.9%)
  Arms: Placebo

SUMMARY:
This is a phase I, prospective, three-arm, open-label, randomized, first in human (FIH) clinical trial to assess the safety and immunogenicity of EgyVax vaccine candidate for prophylaxis of SARS-CoV-2 infection (COVID-19).

DETAILED DESCRIPTION:
Study subjects will receive one dose of study intervention as assigned at each vaccination visit (Visits 1 and 4) via intramuscular (IM) injection in the upper arm approximately 14 days apart. Study interventions should be administered into the deltoid muscle, preferably of the nondominant arm .

Each subject will be assigned to receive either:

* 35 mcg dose for both vaccinations at day 0 and day 14 (low dose, 15 subjects)
* 70 mcg dose for both vaccinations at day 0 and day 14 (high dose, 15 subjects)
* Placebo for both injections at day 0 and day 14 (Placebo, 15 subjects)

For easier reference, refer to the below definitions of each study group:

* Cohort 1: first three subjects of the low dose vaccination group plus two subjects from the control group
* Cohort 2: second three subjects of the low dose vaccination group plus one subject from the control group
* Cohort 3: remaining nine subjects of the low dose vaccination group plus two subjects from the control group
* Cohort 4: first three subjects of the high dose vaccination group plus two subjects from the control group.
* Cohort 5: second three subjects of the high dose vaccination group plus one subject from the control group
* Cohort 6: remaining nine subjects of the high dose vaccination group plus two subjects from the control group

Step 1 (Day 0): Cohort 1 will receive their initial dose of vaccine.

Step 2 (Day 7): After 7 days from step 1, Cohort 2 will receive their initial dose of vaccine.

Step 3 (Day 14): After 7 days from step 2; Cohort 1 will receive their second dose of vaccine, and Cohort 3 & 4 will randomly receive their initial dose of vaccine.

Step 4 (Day 21): After 7 days from step 3, Cohort 2 will receive their second dose of vaccine, and Cohort 5 will receive their initial dose of vaccine

Step 5 (Day 28): After 7 days from step 4, Cohort 3 & 4 will receive their second dose of vaccine, and Cohort 6 will receive their initial dose of vaccine

Step 6 (Day 35): After 7 days from step 5, Cohort 5 will receive their second dose of vaccine

Step 7 (Day 42): After 7 days from step 6, Cohort 6 will receive their second dose of vaccine.

The Data Monitoring Committee (DMC) will periodically review trial data including safety data. Subjects will also be asked to provide blood samples at specified time points, which investigators will test in the laboratory to detect and measure the immune response to the vaccine candidate

ELIGIBILITY:
Inclusion Criteria:

1. Provides proven legal identity.
2. Provides written informed consent prior to initiation of any study procedures.
3. Willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Agrees to the collection of venous blood per protocol.
5. Male or non-pregnant female subjects, 18-55 years of age at the time of enrollment.
6. Male or female of childbearing potential must agree to use or have practiced true abstinence or use at least two acceptable primary form of contraception from first vaccination until 60 days after the last vaccination.
7. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to each vaccination.
8. Healthy subjects who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
9. Oral temperature is less than 37.5 °C.
10. Pulse less than 100 beats per minute.
11. Blood pressure (BP) less than 140/90 mm Hg, inclusive. (Appendix I)
12. Clinical screening laboratory evaluations (white blood cell (WBC), hemoglobin (Hgb), platelets (PLTs), alanine transaminase (ALT), aspartate transaminase (AST), creatinine (Cr), alkaline phosphatase (ALP), total bilirubin (T. Bili), prothrombin time (PT), partial thromboplastin time (PTT) and HbA1c) are within acceptable normal reference ranges at the clinical laboratory being used.
13. Must agree to refrain from donating blood or plasma during the study (outside of this study).

Exclusion Criteria:

1. Positive pregnancy test either at screening or just prior to each vaccine administration.
2. Female subject who is breastfeeding or plans to breastfeed from the time of the first vaccination through 60 days after the last vaccination.
3. Individuals at high risk for severe COVID-19, including those with any of the following risk factors:

   1. Type 1 diabetes (T1D), or type 2 diabetes (T2D) that cannot be controlled by drugs
   2. Hypertension that cannot be controlled by drugs
   3. Current smoking
   4. History of chronic smoking within the prior year
   5. BMI is ≤ 18 kg/m2 or ≥ 40 kg/m2
   6. Resident in a long-term facility
4. Have any other medical disease/condition or psychiatric condition that, in the opinion of the participating site principal investigator (PI) or appropriate sub-investigator, precludes study participation. (Appendix II)
5. History of recent COVID-19 diagnosis; within 6 months prior to enrollment . This should be confirmed with chest computed tomography (CT) scan and or polymerase chain reaction (PCR).
6. Has an acute illness, as determined by the participating site PI or appropriate sub-investigator, with or without fever (oral temperature of 37.8 °C or above) within 72 hours prior to each vaccination. An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
7. Has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) types 1 or 2 antibodies at screening.
8. Has participated in another investigational study involving any investigational product (study drug, biologic or device) within 60 days, or 5 half-lives, whichever is longer, before the first vaccine administration.
9. Currently enrolled in or plans to participate in another clinical study with an investigational agent that will be received during the study-reporting period.
10. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to any previous licensed or unlicensed vaccines.
11. Exposure to radiotherapy or chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness. Including, but not limited to, systemic corticosteroids exceeding ≥20 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar drugs during the preceding 6-month period prior to vaccine administration (Day 0). The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.
12. Anticipating the need for radiotherapy or immunosuppressive treatment within the next 6 months. Including, but not limited to, systemic corticosteroids ≥20 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar drugs during the preceding 6-month period prior to vaccine administration (Day 0). The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.
13. Received immunoglobulins and/or any blood or blood products within the 4 months before the first vaccine administration or at any time during the study.
14. Has any blood dyscrasias or clinically significant disorder of coagulation (in the opinion of the investigator). The use of ≤325 mg of aspirin per day as prophylaxis is permitted, but the use of other platelet aggregation inhibitors, thrombin inhibitors, Factor Xa inhibitors, or warfarin derivatives is exclusionary, regardless of bleeding history.
15. Has any liver disease or impairment, including fatty liver.
16. Has a history of alcohol abuse or other recreational drug use within 6 months before the first vaccine administration.
17. Has a positive test result for drugs of abuse at screening or before the first vaccine administration.
18. Has any abnormality that would interfere with the ability to observe local reactions at the injection site.
19. Received or plans to receive a licensed, live vaccine within 4 weeks before or after each vaccination. For example: Yellow fever, Tuberculosis (BCG), Influenza live attenuated.
20. Received or plans to receive a licensed, inactivated vaccine within 2 weeks before or after each vaccination.
21. Receipt of any other SARS-CoV-2 or other experimental coronavirus vaccine at any time prior to or during the study.
22. Close contact of anyone known to have SARS-CoV-2 infection within 30 days prior to vaccine administration. If exposure is suspected, subjects may be enrolled with subsequent documentation of a negative test for SARS-CoV-2, at the discretion of the investigator.
23. On current treatment with investigational agents for prophylaxis of COVID-19.
24. Currently working in occupations with high risk of exposure to SARS-CoV-2 (e.g., healthcare worker, emergency response personnel).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-02-06 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Safety of EgyVax Vaccine after 1 month from the first vaccination dose | Up to 1 month of the first vaccination dose
  To evaluate the recorded adverse events (AEs) following vaccine administration
Safety of EgyVax Vaccine up to 6 months of the first vaccination dose | Up to 6 months of the first vaccination dose
  To evaluate and follow up the Serious AEs (SAEs) following vaccine administration

SECONDARY OUTCOMES:
Evaluation of Neutralizing antibodies (NAB) response following vaccine administration | Up to 6 month of the first vaccination dose
  To measure the NAB levels following vaccine administration
Dose Selection | After 3 months of the first vaccination dose
  To recommend dose for phase II clinical trials, in terms of safety and NAB response
Safety of EgyVax Vaccine | Up to 1 year of the first vaccination dose
  To evaluate the recorded AEs following vaccine administration

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals (Al-Manial Specialized University Hospital), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. WHO Director-General's opening remarks at the media briefing on COVID-19. Available from: https://www.who.int/dg/speeches/detail/who-director-general-s-opening-remarks-at-the-media-briefing-on-covid-19---11-march-2020 World Health Organization. Coronavirus disease 2019 (COVID-19) situation report - 70. In: Data as reported by national authorities by 10:00 CET 30 March 2020. Geneva, Switzerland: World Health Organization; 2020. Rauch S, Jasny E, Schmidt KE, et al. New vaccine technologies to combat outbreak situations. Front Immunol 2018;9:1963. Saad MA, Saleh AA, Islam Ryan MA, Saleh MS, Abdulaal T, Hassan WA, et al. Preliminary Step towards COVID-19 Inactivated Vaccine Development in Egypt. Archives of Clinical Trials. 2021 Jul 28;1(1). Ali AA, Saad MA, Ryan I, Amin M, Shindy MI, Hassan WA, et al. Safety and Immunogenicity Evaluation of Inactivated whole-virus-SARS-COV-2 In Mice As Emerging Vaccine Development In Egypt. bioRxiv. 2021 Jan 1. US Food and Drug Administration. Guidance for industry: toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials. Rockville, MD: Center for Biologics Evaluation and Research; September 2007. Hobohm L, Becattini C, Ebner M, et al. Definition of tachycardia for risk stratification of pulmonary embolism. European Journal of Internal Medicine. 2020 Dec 1;82:76-82. Williams B, Mancia G, Spiering W, et al. 2018 ESC/ESH Guidelines for the management of arterial hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology (ESC) and the European Society of Hypertension (ESH). European heart journal. 2018 Sep 1;39(33):3021-104.